CLINICAL TRIAL: NCT03728231
Title: Disease Activity in Rheumatoid Arthritis and Systemic Lupus Erythematosus and Its Relation to Muscle Performance,Fatigue and Blood Parameters
Brief Title: Disease Activity in RA and SLE Patients and Its Relation to Muscle Performance,Fatigue and Blood Parameters
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Gamal Seddek, Principle Investigator, Assiut University
Other Study IDs: DAS in RA and SLE
Record Dates: First submitted 2018-10-24; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Diseases | interventions — Blood Cell Count; Immunologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fifty patients with RA.: -CBC with assessment of NLR and PLR. Immumological tests (RF, ANA, anti-ds DNA).
  * Functional Performance Tests:(12)
  * Fatigue severity scale (13).
  * Short-Form Health Survey 36 (SF-36) (14).
  * the short version of the International Physical activity Questionnaire (s-IPAQ) (15).
  * frequency intensity time (FIT) index of kasari (16). :* Disease activity Score(DAS)(17)
  Interventions: Other: Complete blood count
- Fifty patients with SLE.: CBC with assessment of NLR and PLR. Immumological tests (RF, ANA, anti-ds DNA).
  * Functional Performance Tests:(12)
  * Fatigue severity scale (13).
  * Short-Form Health Survey 36 (SF-36) (14).
  * the short version of the International Physical activity Questionnaire (s-IPAQ) (15).
  * frequency intensity time (FIT) index of kasari (16). :* SLE Disease activity Index(SLEDAI)(18)
  Interventions: Other: Complete blood count
- Fifty apparently healthy controls: CBC with assessment of NLR and PLR. Immumological tests (RF, ANA, anti-ds DNA).
  * Functional Performance Tests:(12)
  * Fatigue severity scale (13).
  * Short-Form Health Survey 36 (SF-36) (14).
  * the short version of the International Physical activity Questionnaire (s-IPAQ) (15).
  * frequency intensity time (FIT) index of kasari (16).
  Interventions: Other: Complete blood count

INTERVENTIONS:
Other: Complete blood count — taking blood sample from venous blood
  Other Names: Immunological tests; ESR and CRP

SUMMARY:
Assessment of disease activity in Rheumatoid Arthritis and Systemic lupus patients related to muscle performance, fatigue and blood parameters

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most common inflammatory arthritis, affecting 0.5-1% of the general population world-wide. It is primarily a disease of the joints, but abnormal systemic immune responses are evident and cause a variety of extra-articular manifestations .

Physical inactivity is one of the key mechanisms affecting skeletal muscle mass and body composition, leading to progressive muscle loss and abdominal fat gain . Muscle strength and endurance are determinants of muscle performance. Relatively little is known about how muscle performance relates to RA clinical variables; also muscle performance is not routinely assessed in clinical practice among patients with RA. Decreased muscle strength has negative outcomes in RA, associating with disease activity, radiological damage and disability .Rheumatoid cachexia, including loss of muscle mass and concomitant increase in fat mass with normal or increased body weight , is a common feature in patients with RA. Assessment of inflammation in RA with markers is important to detect long-term outcome. Parameters of hemogram, particularly those including immune system elements, are important in the assessment of different diseases and/or signs. Immune system elements involve the neutrophils, lymphocytes and platelets that have a role in the control of inflammation, while also undergoing changes secondary to inflammation .

Systemic lupus erythematosus (SLE) is a complex autoimmune disease with chronic relapsing-remitting course and variable manifestations varying from mild mucocutaneous to severe, life-threatening illness .

It has been speculated that fatigue, a symptom frequently observed in approximately 80% of SLE patients , may contribute to a reduction in physical fitness (i.e.,muscle weakness and low cardiovascular capacity) which, in turn, leads to an impairment in the performance of activities of daily living and in the overall quality of life .

SLE patients experienced decreased physical function, low dynamic muscle strength capacity, and poor quality of life, suggesting that either "residual" fatigue or other factors (e.g., long-term medication or systemic inflammation) may have contributed to the poor health-related findings .

Celikbilek et al. observed that Neutrophil /Lymphocyte Ratio (NLR) and Platelet/Lymphocyte Ratio (PLR) in peripheral blood are simple Systemic Inflammatory Response (SIR) markers which are evaluated by blood parameters and showed that NLR possesses a diagnostic value in certain pathologies characterized by systemic or local inflammatory response. Amaylia et al. found that NLR was significantly higher in SLE than normal subjects .

ELIGIBILITY:
Inclusion Criteria::

1. RA diagnosis according to 1987ACR criteria,or 2010 ACR/EULAR criteria
2. SLE diagnosis according to 1982 ACRor 2012 ACRcriteria
3. Patients aged > 18 years.
4. Stable disease with no activity during last 3 months.
5. Regular medication in last 3 months.

Exclusion Criteria:

1. Subjects with hematologic disorders other than anaemia.
2. Concomitant infectious or inflammatory diseases such as ulcerative colitis.
3. Liver or kidney disease.
4. Coronary heart disease.
5. Other immunological diseases.
6. Pregnant ladies.
7. Patients with end stage organ failure.
8. Patients with malignancies.
9. Patients receiving any medications affect blood picture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty patients diagnosed Rheumatoid arthritis according to 1987ACR or 2010ACR\EULAR criteria Fifty patients diagnosed Systemic lupus according to 1982 ACRor 2012ACR criteria Fifty Apperantly healthy persons
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-11-11 (Estimated); Study Completion 2020-02-02 (Estimated)

PRIMARY OUTCOMES:
estimation of muscle performance in Rheumatoid arthritis and Systemic lupus patients by 30_s chair stand test (repetition 4_12) . | 6 months
  use of 30_s chair stand test(repetition 4_12) in detection of degree of muscle performance in Rheumatoid arthritis and Systemic lupus patients .

REFERENCES:
- [Background] Biolo G, Cederholm T, Muscaritoli M. Muscle contractile and metabolic dysfunction is a common feature of sarcopenia of aging and chronic diseases: from sarcopenic obesity to cachexia. Clin Nutr. 2014 Oct;33(5):737-48. doi: 10.1016/j.clnu.2014.03.007. Epub 2014 Mar 29. PMID 24785098
- [Background] Hakkinen A, Kautiainen H, Hannonen P, Ylinen J, Makinen H, Sokka T. Muscle strength, pain, and disease activity explain individual subdimensions of the Health Assessment Questionnaire disability index, especially in women with rheumatoid arthritis. Ann Rheum Dis. 2006 Jan;65(1):30-4. doi: 10.1136/ard.2004.034769. Epub 2005 May 18. PMID 15901635
- [Background] Summers GD, Metsios GS, Stavropoulos-Kalinoglou A, Kitas GD. Rheumatoid cachexia and cardiovascular disease. Nat Rev Rheumatol. 2010 Aug;6(8):445-51. doi: 10.1038/nrrheum.2010.105. Epub 2010 Jul 20. PMID 20647995
- [Background] Alaranta H, Hurri H, Heliovaara M, Soukka A, Harju R. Non-dynamometric trunk performance tests: reliability and normative data. Scand J Rehabil Med. 1994 Dec;26(4):211-5. PMID 7878396
- See also: 9.Balsamo et al. BMC MusculoskeletalDisorders 2013, 14:263 — http://www.biomedcentral.com/1471-2474/14/263
- See also: 2.Biolo G, Cederholm T, Muscaritoli M. Muscle contractile and metabolic dysfunction isacommonfeature ofsarcopenia of ang and chronic diseases: From sarcopenic obesity to sarcopenic obesity to cachexia. Clin Nutr. 2014; 33:737-748 — https://doi.org